CLINICAL TRIAL: NCT05052775
Title: EFFICACY OF MORUS ALBA FRUIT EXTRACTS AND CHLORHEXIDINE ON SALIVARY STREPTOCOCCUS MUTANS AND pH LEVELS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Eid Muhammad, M.Phil Trainee, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2380720EMOM
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries
Keywords: Dental Caries; Chlorhexidine; Morus Alba
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Masking Description: Total number of groups = 3 Group 1 has been given chlorhexidine mouthwash and group 2nd and 3rd have been given 20% and 30% aqueous extract of morus alba fruit respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chlorhexidine Group (Active Comparator): These patients were control group given chlorhexidine mouthwash 2 times per day for 15 days
  Interventions: Other: Chlorhexidine Mouthwash
- Morus Alba 20% (Experimental): Patients were given morus alba 20% concentration 2 times per day for 15 days
  Interventions: Other: Morus Alba 20%
- Morus Alba 30% (Experimental): Patients were given morus alba 30% concentration 2 times per day for 15 days
  Interventions: Other: Morus Alba 30%

INTERVENTIONS:
Other: Chlorhexidine Mouthwash — Patients were given chlorhexidine mouthwash 2 times per day for 15 days
  Arms: Chlorhexidine Group
Other: Morus Alba 20% — Patients were given morus alba 20% concentration 2 times per day for 15 days
  Arms: Morus Alba 20%
Other: Morus Alba 30% — Patients were given morus alba 30% concentration 2 times per day for 15 days
  Arms: Morus Alba 30%

SUMMARY:
Dental caries is highly prevalent across the globe including Pakistan and is associated with tooth loss, malocclusion and temporomandibular joint problems and sometimes may cause life threatening infections. Streptococcus mutans is considered to be one of the major pathogen responsible for the development of dental caries. As treatment of dental carries is quite expensive, main focus is on the prevention of dental carries. Chlorhexidine is the gold standard mouthwash used for the prevention of dental carries but its use has been associated with certain side effects including staining of teeth, burning sensation and a bitter taste in the oral cavity. Many populations use medicinal plants as traditional or alternative treatments for various ailments due to their better safety profiles, health beneficial effects, lower cost and easy availability. Among the plant species used for medicinal purposes are those of the genus Morus. Its most commonly used species are Morus alba, rubra and nigra that have also shown antimicrobial properties against various infections in addition to other health promoting effects. Moreover, morus alba fruit has not been evaluated for its antimicrobial activity against oral pathogens including streptococcus mutans. The purpose of this study is to evaluate the antimicrobial properties against salivary streptococcus mutans and alteration of pH in the saliva of patients with dental caries before and after the use of chlorhexidine and morus alba fruit extract mouthwashes.

This study is double blinded randomised clinical trial. Sample size is calculated according to open Epi calculator and came out as 1 in each group. We will take sample size as 120 and the sampling technique will be non-probability consecutive sampling. Morus alba extract preparation will be done in the Botany department of Lasbella University of Agriculture, Water and Marine Sciences (LUAWMS) Balochistan. According to inclusion criteria and after obtaining informed consents, samples of saliva of the individuals of 18-40 year of both genders will be collected from the OPD of Dentistry department, Civil hospital Uthal Balochistan at the beginning of the study and two weeks after the treatments. The total 120 subjects will be equally divided into three groups, 40 participants in each group (A, B and C). The subjects in group A will be given chlorhexidine mouthwash and the subjects in group B and C will be given 20% and 30% aqueous extracts of morus alba fruit in the form of mouthwashes respectively. The samples of saliva will be analysed for S.mutans counts and pH levels at baseline and 15 days after the use of respective mouthwash. Culture procedure for S.mutans count will be Dilution and Spread plate technique.

DETAILED DESCRIPTION:
INTRODUCTION Streptococcus mutans is the major pathogen involved in the development of dental caries. This is an anaerobic gram positive coccus, naturally present in the oral microbiota and can easily colonize on the tooth surface and initiates production of acid by combining extracellular polysaccharide that results in demineralization of tooth and development of dental caries (Shah et al., 2018). The quantity of colonized surfaces is associated with streptococcus mutans in the saliva. Thus, by decreasing the concentration of Streptococcus mutans in the mouth cavity would have a significant advantage in reducing the occurrence of cariogenic microbes. (Lemos et al., 2019, Forssten et al., 2010, Banas and Drake., 2018) Dental caries is a microbial disease of the oral cavity, which is identified by demineralization of the inorganic substances and dissolution of the organic substances of the teeth. Dental caries has been recognized throughout history and exists around the world, reported to be 44%, but the severity and prevalence changes in different countries (J.V Soames and J.C Southam et al., 2018). In our neighboring countries, the frequency of dental caries is quite high, documented to be 68%, 65% and 64% in China, Iran and India respectively. The prevalence of dental caries in Pakistan is also quite high, around 62%, which is associated with significant morbidity and economic consequences (Reddy K S, et al., 2017, Lu Liu et al., 2013) Dental caries basically involves contact between the tooth structure, the sugars and biofilm formed on the tooth surfaces (Pitts, N. B et al., 2016). The caries process composed of altering periods of demineralization and remineralization of tooth, which, if net demineralization happens over adequate time, results in the initiation of dental caries. The cause of dental caries is lactic acid produced by fermentation of sugars by oral bacteria (Banas and Drake., 2018). The normal pH level of saliva is 6.2- 7.6. At neutral pH, calcium and phosphate ions from the saliva incorporate into the enamel and maintain the structure of enamel, but when the pH level falls below normal, i.e. at 5.5 or below 5.5, the calcium and phosphate ions from the enamel leach out and causes the exchange of minerals ions from hydroxyapatite crystals of enamel into plaque, resulting in demineralization of tooth (J.V Soames Oral pathology 2018).

Dental caries management emphasizes on reducing tooth demineralization by changing eating habits, altering or inhibiting bacterial growth, changing the salivary pH level and buffering capacity (Khirtika et al., 2017, Velmurugan et al., 2013, Yang et al., 2018). Different antimicrobial synthetic mouthwashes, toothpastes, gels, chewing gums and varnishes have been used to improve mouth hygiene and prevent dental caries by aiming cariogenic microorganisms. The prevention of dental caries is done by mouth brushing after meal, by using fluoride toothpastes, antimicrobial mouthwashes, interdental cleaning aids, salivary stimulants (xylitol, mannitol), pit and fissure sealants, and application of topical fluoride on teeth surfaces. Mouth rinses also reduce gingival inflammation and inhibit plaque formation (Velmurugan et al., 2013, Chen and Wang, 2010, Zajkani et al., 2018). Mouthwashes have anticariogenic effects, but have certain disadvantages. They are costly, have side effects including staining of the teeth and burning sensation in the oral cavity (Nayak et al., 2012, Aoun et al., 2018).

Chlorhexidine is gold standard, commonly used and most effective chemical approach to decrease the accumulation of plaque. Daily rinsing mouth with chlorhexidine (0.2%) has been shown to reduce the growth rate of streptococcus mutans in the oral cavity (Velmurugan et al., 2013). However, it has certain side effects, i.e. oral mucosal erosion, parotid swelling, staining of teeth, burning feeling and bitter taste. (Jacob and Nivedhitha, 2018b, Shah et al., 2018, Van der Weijden et al., 2010, Nayak et al., 2012, Solderer et al., 2019) Many populations use medicinal plants as traditional or alternative treatments for various ailments due to their better safety profiles, health beneficial effects, lower cost and easy availability. Among the plant species used for medicinal purposes are those of the genus Morus, includes most commonly used species are Morus alba, rubra and nigra, that have also shown antimicrobial properties against various life threatening infections (Ercisli S et al., 2006). Morus alba commonly called as white mulberry, and it belongs to family Moraceae is otherwise called Tut, shahtoot or mulberry. Morus Alba (white mulberry) is native to China, India, Pakistan and Japan (Kumar V et al., 2008). In the current study, Morus alba fruit extract will be compared with chlorhexidine to Streptococcus mutans against oral pathogens due to its antimicrobial properties.

Statement of the problem Dental caries is highly prevalent across the globe including Pakistan; it causes tooth loss, malocclusion, and temporomandibular joint problems. The associated infections may carry risk of spreading into superficial and deep fascial spaces and, even may cause life threatening infections. Treatment of dental caries is quite expensive and poses an economic burden on our already deprived low socioeconomic population. So, there is need of exploration of natural products that may have antimicrobial and other beneficial effects to decrease the caries activity along with good safety profiles, easily available and cost-effective.

Research question Are the aqueous extracts of Morus alba fruit equally effective as chlorhexidine mouthwash for the prevention of dental caries? Objectives To compare the efficacy of Morus alba fruit extracts with chlorhexidine in patients having dental caries on the basis of reduction in counts of Streptococcus mutans in their saliva.

To compare the efficacy of Morus alba fruit extracts with chlorhexidine in patients having dental caries on the basis of increase in their salivary pH levels.

Rationale Chlorhexidine is a chemical, having bitter taste and cause burning sensation in the oral cavity and may not be feasible for the patients due to cosmetic reasons. Mouthwash derived from herbal products, having antimicrobial activity against oral pathogens might provide economical and safe treatment option to reduce the burden of dental caries in our clinical set-up. To the best of our knowledge, the mulberry fruit extract has not been evaluated for its antimicrobial activity against oral pathogens including Streptococcus mutans.

Hypothesis

Null hypothesis:

Ho: Aqueous extracts of Morus alba fruit are not equally effective as chlorhexidine mouthwash for the prevention of dental caries.

Alternate Hypothesis:

Ha: Aqueous extracts of Morus alba fruit are equally effective as chlorhexidine mouthwash for the prevention of dental caries.

REVIEW OF LITERATURE Dental caries consists of connections between the tooth structures, sugars, and the microbial biofilm on the tooth surfaces (Pitts, N. B et al., 2016). Streptococcus mutans and salivary pH are the two main factors that cause dental caries and therefore targeting them can be an efficient route to tackle this global disease. Chlorhexidine is an excellent antimicrobial agent and considered as boon for maintaining oral health and hygiene. Similarly, many herbal agents has been introduced which are as effective as chlorhexidine. (Sajjan et al., 2016, Ahmed et al., 2017, Jacob and Nivedhitha, 2018, Carounanidy et al., 2007, Esther et al., 2017) Medicinal plants have been used by many populations as a therapeutic agent because of their easy availability, safe and cost effectiveness. The morus species also have medicinal properties and have been used as antidiabetic, neuroprotective, hypolipidimic and as laxatives (Anna Gryn-Rynko et al., 2016). More than 100 species of morus are present all over the world and in Pakistan there are 25 morus species available. The most common morus species are Morus alba, rubra and nigra (Imran M., Khan H., et al., 2010).

Morus alba fruit contains many active substances, such as flavonols, polyphenols, alkaloids and polysaccharides (Gundogdu M et al., 2011). Morus alba is the rich source of Vitamin A, Vitamin B1, Folic acid, Vitamin C, Minerals, Carbohydrates, Amino acids, Fatty acids, anthocyanin and saponins (Jiang Y et al., 2015).

In conventional Chinese natural medication, mulberry fruit have been utilized in people drugs to treat diabetes, hypertension, anemia, and joint pain. Morus alba has been known for its antidiabetic, antihelmintic, antimicrobial, anxiolytic, hepatoprotective and nephroprotective properties (Wang, J.; et al., 2013, Yang, X. L et al., 2010, Khalid, S et al., 2017). The Morus fruit, although from the same species, that may contain different antioxidant properties as well as different chemical composition. The mineral elements in Morus alba include potassium (K), sodium (Na), phosphorus (P), calcium (Ca), zinc (Zn), iron (Fe), copper (Cu), manganese (Mn), selenium (Se), magnesium (Mg), chromium (Cr), and arsenic (As) (Liang, L et al., 2012).

The methanolic extract of the bark of Morus alba and its constituents are used as antimicrobial agents (Kuete, et al., 2009). The antimicrobial agent "kuwanon G" obtained from bark of the root of Morus alba has indicated activity against Streptococcus mutans at a MIC of 8.0 μg/ml. The bactericidal test of kuwanon G indicated that it totally inactivated Streptococcus mutans at the concentration 20 μg/ml in 60 seconds (Park, K. M et al., 2002).

According to Jha et al, he assessed the antimicrobial activity of Morus alba leaves (aqueous extract) on gram positive (Staphylococcus aureus, Bacillus subtilis), and gram negative bacteria (Pseudomonas aeruginosa and Escherichia coli). Results of the antimicrobial activity confirmed that Bacillus subtilis, Pseudomonas aeruginosa, Staphylococcus aureus and Escherichia coli were most susceptible bacterial species to crude extract, showed the MIC value at concentration from 0.2-26mg/mL (S. Jha, A.K et al., 2013).

The antimicrobial activity of 1-deoxynojirmiycin (component of Morus alba leaves) and crude ethanolic extract of Morus alba leaves were assessed. Both the 1-deoxynojirmiycin and morus alba leaves (crude extract) showed strong bacteriostatic activity against Streptococcus mutans, but the 1-deoxynojirmiycin showed lower MIC value (15.6mg/ml) than the crude extract of Morus alba (125mg/mg/mL) ( B. Islam., et al 2008). The ethanolic extract of Morus alba leaves showed antimicrobial activity against Pseudomonas aeruginosa, Staphylococcus aureus, Candida krusei, Candida albicans, Aspergillus flavus and Candida tropicalis (Oliveira et al., 2015).

Anthocyanins are the most significant constituent of Morus alba fruit, which are phenolic compounds that are responsible for many biological activities such as antimicrobial, antioxidant, neuroprotective, and anti-inflammatory properties (Liu LK et al., 2008). The cyanidin-3-glucoside and cyanidin-3-rutinoside are the main anthocyanins separated from mulberry fruit (Suh H.J et al 2003, Liu X.et al 2004). The active ingredient of Morus alba is anthocyanin and anthocyanin present in the fruit of Morus species displayed antibacterial activities against E. coli, Pseudomonas aeruginosa, and Staphylococcus aureus (Chen H., et al 2017). The proposed mechanisms by which anthocyanin produces antimicrobial effects include action on the cell membrane of pathogen with the leakage of its nucleic acid and proteins (Bajpai et al., 2013). Anthocyanin causes inhibition of microbial superoxide dismutase, alkaline phosphatase and ATP production with subsequent inhibition of TCA cycle (Li et al., 2010).All these mechanisms results in the lysis of pathogenic cell.

Shumaila Naz et al confirmed the antimicrobial activity of Mulberry fruit extracts against water- borne microbial pathogens (Listeria monocytogene, Salmonella enteric, Moraxella catarrhalis, Legionella pneumophila, Micrococcus luteus, Proteus mirabilis, Clostridium sp., Serratia sp., Aeromonas hydrophila , Corneybacterium sp., Bacillus subtilis, , E. coli, Bacillus megaterium, Bacillus thuringiensis, Streptococcus pyogenes, Actinomyces sp., Staphylococcus aureus, Vibrio cholera, Salmonella typhi, Bacillus anthracis and Streptococcus pneumonia) isolated from different water samples. The results indicated that mulberry fruit extracts are effective against water-borne microbial pathogens (Shumaila Naz et al., 2018).

SAFETY PROFILES OF MORUS ALBA The intragastric administration of Morus alba extract in rats for the duration of 7 days at the maximum dose of 1gm/kg didn't produce toxic effects (Jiao Y et al., 2017). A study conducted on rats in which the effects of ethanolic extracts of Morus alba in rats at the dose of 250mg/kg for 2 weeks of administration did not cause toxic effects (Hwang et al., 2016). Another study conducted on rats that were fed with anthocyanins derived from mulberry fruit. The anthocyanins decreased the raised levels aspartate aminotransferase (AST) and alanine aminotransferase ALT in rats. (Hepatoprotective effects) SAMPLE SIZE CALCULATION The sample size was estimated using Open Epi sample size calculator by considering the following statistics; Change in pH level (Chlorhexidine) = 6.88±0.20 (Velmurugan et al., 2013) and considering 20% difference in pH for mulberry extracts as 8.256±0.24 Power of test= 90% Confidence level= 95% The calculated sample size came out as 1 in each group. However, I will include 120 patients having 40 patients in each group according to normality assumption.

RESEARCH METHODOLOGY Study setting This study will be conducted at the department of Dentistry, Civil hospital Uthal, district Lasbella and at the department of Plant Pathology, Lasbella University of Agriculture, Water and Marines Sciences (LUAWMS) Balochistan.

Study design Randomized Controlled Clinical Trial It's a double blinded study, in which both researcher and the patient will be blinded to keep the results unbiased. However, the co-investigator will know either the patient is receiving gold standard or herbal mouthwash.

Study duration The study duration will be of 6 months to 1 year after approval of study from RAC, ERC and BASR of Ziauddin University.

Sampling technique Non-Probability consecutive sampling technique will be employed for the sample selection

Selection criteria Inclusion criteria All the patients of age 18-40 years at least 20 teeth in their mouth and not including wisdom teeth.

The patients of either gender. The patients with active and untreated carious lesions, (at least one carious tooth should be present in patient oral cavity).

Exclusion criteria The patients undergoing orthodontic treatment The patients already taking antibiotic therapy or antimicrobial rinse. The patients having allergy to chlorhexidine mouthwash The patients whose consents could not be obtained MATERIALS AND METHOD MATERIALS USED IN STUDY The materials used in the study will be Chlorhexidine mouthwash, Morus alba fruit, pH meter, selective agar and culture plates for Streptococcus mutans, test tubes and saliva collections kits.

MORUS ALBA COLLECTION Morus alba (White Mulberry) fruit will be obtained from an authentic herbal store and the Morus alba fruit will be authenticated from Botany department of LUAWMS.

PREPARATION OF AQUEOUS EXTRACT OF MORUS ALBA FRUIT The preparation will be done in the department of Plant Pathology LUAWMS. Morus alba fruit will be washed with distilled water and will be allowed to dry. Then the fruit material (Morus alba) will be grinded with help of mortar and pestle. For 20% aqueous preparation, 100ml distilled water will be added to 20g grinded powder and will be incubated in shaking incubator for 8 hours. (For 30% aqueous preparation, 100ml distilled water will be added to 30g grinded powder). Aqueous extracts will be filtered through Watman No. 1 (Schuell and Schleicher 125 mm Cat No. 1001 125) filter paper (Shumaila naz et al., 2018).

STANDARDIZATION OF PARTICIPANTS The subjects selected according to inclusion criteria will be standardized. The participants will be advised to brush their teeth twice a day (after breakfast in the morning and at bed time), and to avoid junk foods. Participants will be advised to take sugary drinks (tea, coffee, sweetened beverage) not more than 2 times a day. These Instructions will also be given to participants in written form. The participants will be instructed to act upon this guidance and will be called after 1 week for baseline salivary samples.

DATA COLLECTION PROCEDURE A total of 120 patients fulfilling the inclusion criteria will be enrolled in the study. Informed consents will be taken from all the participants. While taking consent, the patients will be informed that they will receive either gold standard (chlorhexidine) or herbal mouthwash. The selection of patients either in group A, B or C will be done by Random Number Table method. The labeling of group as A, B and C will be done by co-investigator. List of groups will be sealed in opaque envelop and will opened when study will be completed.

STUDY GROUPS A total of 120 participants will be included in the study. The participants will be equally divided into three groups (group A, B and C). The participants in group A will be given Chlorhexidine mouthwash and the participants in the group B and C will be given 20% and 30% aqueous extract of Morus alba fruit respectively.

SALIVARY pH ANALYSIS The salivary pH level analysis will be done using pH meter and the salivary pH will be recorded at baseline and 15 days after the use of respective mouthwash.

EXPERIMENTAL PROCEDURE The 5ml baseline unstimulated salivary samples will be taken from the participants by Passive drooling technique, then 3ml will be used for measurement of salivary pH and the remaining salivary sample will be stored at 0 C, and then will be transferred to lab for the assessment of Streptococcus mutans. After baseline salivary samples taken, participants will be asked to rinse and hold 10ml of respective mouthwash for the duration of 30 seconds in their mouth before spitting it. The procedure will be repeated by the participants, twice a day for 15 days. After 15 days, salivary samples will be taken again from participants for assessment of Streptococcus mutans and the results obtained will be compared with baseline salivary samples for Streptococcus mutans.

CULTURE PROCEDURE The technique for assessing the microbial content will be dilution and spread plate method. Salivary microbial analysis will be done by diluting each salivary sample 1:10 ratio in distilled water. Each sample will be then streak into plate having Mitis salivarius agar media (MSA). Plates will be then incubated for 48 hours at 37°C and the number of Streptococcus mutans colonies (CFU) will be counted under self-illuminating binocular microscope. All findings will be recorded in pre-designed proforma. (Smariti sexena et al,. 2017, Velmurugan et al,. 2013, Hongkun Wu et al., 2003) STATISTICAL ANALYSIS Data will be analyzed using SPSS version 23. Mean and Standard deviation will be taken for numerical data. Frequency and percentages will be taken for categorical data.

Paired-t test will be done for comparison between pre and post intervention values of bacterial counts and pH values for each group and the ANOVA with post hoc Tukey's test will be applied for comparison between three groups. P < 0.05 will be considered as statistically significant.

ETHICAL CONSIDERATION Ethical approval will be taken from the Ethics Committee of Ziauddin University. Informed Consent will be obtained from each subject before recording of any measurement. All information gathered from the study will be kept strictly confidential. Anonymity of all subjects will be maintained by careful storage of information. If any dental related problems will be noticed, then the patients will be informed and referred to the relevant clinics for necessary treatment.

SIGNIFICANCE OF THE STUDY If the results of our study prove Morus alba to be more effective, then being derived from natural source, a safe , low cost and eco-friendly agent will be available in future for the prevention of dental caries. The Morus alba also could be used for children and those who cannot use synthetic mouthwashes due to irritation, alteration of taste, burning sensation and for cosmetic reasons.

Morus alba like other herbal product is eco-friendly and its formulation as an antimicrobial oral rinse helps to minimize the toxic effects on environment produced by chemically produced oral rinse chlorhexidine, which is currently the gold standard agent for dental carries. The results of this study may open doors for other researches on other herbal products traditionally used for their antimicrobial potential.

ELIGIBILITY:
Inclusion Criteria:

All the patients of age 18-40 years at least 20 teeth in their mouth and not including wisdom teeth.

The patients of either gender. The patients with active and untreated carious lesions, (at least one carious tooth should be present in patient oral cavity).

-

Exclusion Criteria:

The patients undergoing orthodontic treatment The patients already taking antibiotic therapy or antimicrobial rinse. The patients having allergy to chlorhexidine mouthwash The patients whose consents could not be obtained

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
count of bacteria (streptococcus mutans)will be decrease | 15 days
  streptococcus mutans is the dental caries causing microorganism, in this study, the count of streptococcus mutans is measured before and after the use of respective mouthwash,the bacterial count decrease after the use of mouthwash, so primary outcome is that there is less chance of dental caries after use of respective mouthwash

CONTACTS AND LOCATIONS:
Overall Officials: Eid Muhammad, MPHIL, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan